CLINICAL TRIAL: NCT03136562
Title: Prevalence of Adrenal Insufficiency in Kidney Transplanted Patients (NTx) in Glucocorticoid Treatment
Brief Title: Prevalence of Adrenal Insufficiency in Kidney Transplanted Patients in Glucocorticoid Treatment
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor, MD, DMSc, Rigshospitalet, Denmark
Other Study IDs: NTx-CSI
Record Dates: First submitted 2017-02-21; First posted 2017-05-02 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood and saliva.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney transplanted patients: Kidney transplanted patients in prednisolone treatment. Adrenal function is assessed by a synacthen test.
  Interventions: Diagnostic Test: Synacthen test
- Control group: Patients in dialysis not in prednisolone treatment. Adrenal function is assessed by a synacthen test.
  Interventions: Diagnostic Test: Synacthen test

INTERVENTIONS:
Diagnostic Test: Synacthen test — 250 microg synacthen test performed fasting, in the morning. P-cortisol measured before and 30 minutes after Synacthen injection.

SUMMARY:
The primary purpose of this study is to determine the prevalence of adrenal insufficiency in a population of patients with kidney transplants receiving low dose prednisone treatment.

Development of glucocorticoid-induced adrenal insufficiency is a serious adverse effect to glucocorticoid treatment. The study includes a control group of patients with kidney failure currently treated in dialysis, who are not in glucocorticoid treatment.

Individual genotyping is performed to determine the haplotype of glucocorticoid receptor polymorphisms: N363 S, BclI, ER23/23EK and 9β in all the patients with the purpose of investigating this as a risk factor for the development of adrenal insufficiency. The hypothesis is that subjects with one or another of the polymorphisms in the glucocorticoid receptor gene will either have increased or diminished glucocorticoid sensitivity.

Using validated questionnaires assessing the quality of life and functional level of the patients enrolled in the study we aim to establish a link between functional level and biochemically proven adrenal insufficiency.

Other secondary outcomes in the study includes bloodpressure, body composition, bone density, metabolic syndrome, inflammation and salivary cortisol profiles.

DETAILED DESCRIPTION:
Adrenal function is assessed in 30 prednisolon treated kidney transplanted patients and compared with 30 patients in dialysis, who are not treated with glucocorticoids. Adrenal function is evaluated using a 250µg Synacthen® test, performed fasting, in the morning, 48 h after the last prednisolone dose.

Cut-off for normal adrenal function is locally validated assay specific cut-off of 30 min P-cortisol >420 nmol/l. The primary outcome measure of this study is P-cortisol concentrations 30 minutes after Synacthen® injection in prednisolone treated patients compared with comtrols. Secondary, 30 minutes P-cortisol is examined in relation to glucocorticoid receptor haplotypes.

The genotyping is determined using polymerase chain reaction (PCR).

The questionnaires used in this study includes EQ-5D, SF-36, Patient Life Situation Form, CushingQol and ADDOQol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years).
* Kidney transplated patients or patients with kidney failure treated in dialysis.
* Prednisone min 5 mg/day max 7,5 mg/day for the kidney transplanted patients (control group not treated with prednisone).

Exclusion Criteria:

* Other major organ disease.
* Anemia with hemoglobin level less than 6,5 mmol/L.
* Not willing to pause any oestrogen tratment for a minimum of 6 weeks.
* Pregnancy.
* Not understanding Danish language or otherwise not able to provide a written informed concent.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 30 kidney transplanted patients and 30 patients in dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of this study is the result of the Synacthen® test using primarily the level of P-cortisol 30 minutes after the injection of synacthen. | The time frame of each Synacthen® test is approximately 90 minutes.
  Cutoff for normal adrenal function: 30 min p-cortisol >/= 420 nmol/L.

SECONDARY OUTCOMES:
Registration of history of treatment. | The registration will take place at the study visit (approximately 90 minutes).
  History of treatment with prednisone and other types of glucocorticoids to examine dosage and time of treatment as risk factors.
Quality of life and functional level. | Patients receive and fill out the questionnaires prior to their arrival at the study visit and hand them in after the Synacthen® test. Patients receive questionnaires either by mail or at one of their visits in the out patient clinic.
  Assessed in all patients enrolled in the study using validated questionnaires as a means to establish a link between functional level and biochemically proven adrenal insufficiency.
Determination of the specific type of glucocorticoid receptor using genotyping in all the patients with the purpose of investigating this as a risk factor for the development of adrenal insufficiency. | Blood for genotyping is sampled from each patient at the study visit during the Synacthen® test. The blood samples are stored frozen and analyzed concurrently.
  Patients are genotyped for 4 polymorphisms (9 beta, ER22/23EK, Bcl1 and N363S) of the glucocorticoid receptor.
Body composition | After the Synacthen® test the height, weight, waist and hip circumference are measured at the study visit.
  Height, weight, waist and hip circumference.
Bone density. | The results from latest Dxa-scan performed in rutine settings are collected from the patients on the same day as the Synacthen® test.
  Results from Dxa-scan.
Metabolic syndrome. | The waistline and blood pressure are measured at the study visit after the Synacthen® test. The blood samples are collected as part of the test and analyazed on the same day.
  Waistline, triglyceride level, HDL cholesterol level, blood pressure and fasting blood sugar is assessed in all the patients.
Salivary cortisol profiles. | Saliva is sampled from each patient at the study visit as part of the Synacthen® test. The samples are stored frozen and analyzed concurrently after all 60 Synacthen® tests have been performed.
  Cortisol concentration in saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, Professor, Principal Investigator — Department of Endocrinology, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided